CLINICAL TRIAL: NCT02438202
Title: Electroconvulsive Therapy for Treatment of Alzheimer´s Disease
Acronym: ECTAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECTAD
Record Dates: First submitted 2015-04-29; First posted 2015-05-08 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electroconvulsive Therapy (ECT) (Experimental): A modified Electroconvulsive Therapy Series in Patients with Alzheimer's Disease. Device for the intervention ECT will be the Thymatron IV device (Somatics, LLC. Lake Bluff, Illinois, USA).
  Interventions: Device: Thymatron IV device (Somatics)

INTERVENTIONS:
Device: Thymatron IV device (Somatics) — Patients will be treated with a modified routine ECT/maintenance ECT series.

SUMMARY:
Electroconvulsive therapy (ECT) induces a cerebral seizure by electrical stimulation under general anesthesia and muscle relaxation, is regarded as a highly efficient (for specific and severe psychiatric disorders) and extremely safe modern treatment option.

Alzheimer´s disease (AD) is a neurodegenerative disorder which is characterized by progressive cognitive deterioration accompanied by declining activities of daily living, by a variety of behavioral disturbances and by neuropsychiatric symptoms. The clinical progression of disease can be delayed by pharmaceutical therapies like acetylcholinesterase inhibition (e.g. rivastigmine) for 6 to 12 months at most.

Along with the well-known biomarkers of AD (Aß- and tau-proteins) a lower brain-derived neurotrophic factor (BDNF) level is since recently being considered as a negative predictor for the further disease course. In animal experimental studies it was possible to arrest the disease progression with the aid of neurotrophic substances. Many single studies, but also a number of meta-analyses show primary gray matter atrophy in hippocampal, parahippocampal and medial temporal brain regions.

Strikingly, ECT yields exact opposite effects to those caused by AD: an ECT series leads to an increase of serum BDNF-levels in patients. Parallel to this observation evidence exists for gray matter volume gain after an ECT series, especially for the hippocampus.

There is sufficient clinical experience regarding the use of ECT in AD-patients, mainly on the basis of following indications: a) affective disorders and b) behavioral disturbances. A positive effect of ECT on the symptoms of agitation and aggression was assessed in AD patients alongside with a very good tolerability.

To investigate the potential salutary effects of ECT on AD the investigators designed a pilot study with the following concept: Patients with a confirmed AD diagnosis and preexisting stable antidementia medication over at least 6 months will receive a modified maintenance ECT over a total of 27 weeks.

In the proposed pilot study, the investigators hypothesize that cognitive functioning of AD patients will improve significantly and independently from affective symptoms, when initial and final examinations are compared. The affirmation of the hypothesis would provide not only further insight into the mechanism of action of ECT but also a very important reference point for the development of new treatment options for a so-far incurable disease.

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) induces a cerebral seizure by electrical stimulation under general anesthesia and muscle relaxation, is regarded as a highly efficient (for specific and severe psychiatric disorders) and extremely safe modern treatment option.

Alzheimer´s disease (AD) is a neurodegenerative disorder which is characterized by progressive cognitive deterioration accompanied by declining activities of daily living, by a variety of behavioral disturbances and by neuropsychiatric symptoms. All currently available treatments remain palliative in nature. The clinical progression of disease can be delayed by pharmaceutical therapies like acetylcholinesterase inhibition (e.g. rivastigmine) for 6 to 12 months at most.

Along with the well-known biomarkers of AD (Aß- and tau-proteins) a lower brain-derived neurotrophic factor (BDNF) level is since recently being considered as a negative predictor for the further disease course. In animal experimental studies it was possible to arrest the disease progression with the aid of neurotrophic substances. Many single studies, but also a number of meta-analyses show primary gray matter atrophy in hippocampal, parahippocampal and medial temporal brain regions.

Strikingly, ECT yields exact opposite effects to those caused by AD: an ECT series leads to an increase of serum BDNF-levels in patients. Parallel to this observation evidence exists for gray matter volume gain after an ECT series, especially for the hippocampus.

There is sufficient clinical experience regarding the use of ECT in AD-patients, mainly on the basis of following indications: a) affective disorders and b) behavioral disturbances. A positive effect of ECT on the symptoms of agitation and aggression was assessed in AD patients alongside with a very good tolerability. A recent review on ECT treatment in patients with concomitant depression and AD pointed out that these patients have significantly better scores in cognitive tests 6 months after the ECT series.

ECT as a psychiatric treatment for cognitive enhancement in AD is uncharted scientific territory.

To investigate the potential salutary effects of ECT on AD the investigators designed a pilot study with the following concept: Patients with a confirmed AD diagnosis and preexisting stable antidementia medication over at least 6 months will receive a modified maintenance ECT over a total of 27 weeks.

In the proposed pilot study, the investigators hypothesize that cognitive functioning of AD patients will improve significantly and independently from affective symptoms, when initial and final examinations are compared. The affirmation of the hypothesis would provide not only further insight into the mechanism of action of ECT but also a very important reference point for the development of new treatment options for a so-far incurable disease.

ELIGIBILITY:
Inclusion Criteria:

* confirmed Diagnostic and Statistical Manual of Mental Disorders (DSM IV) diagnosis of Alzheimer's disease (Mini Mental State Examination >5 and <26)
* routine treatment of AD due to German national guidelines ("S3-Leitlinie")
* Ability to consent. If in doubt an independent (from the study) psychiatrist has to document ability to consent. If no ability to consent is stated, a legal guardian can consent instead. No ECT will be performed against the patient's will.

Exclusion Criteria:

* contraindications for ECT
* current major depressive episode due to DSM IV

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in Cognition | 27 weeks
  individual change between initial and final MiniMentalStateExamination (MMSE)

SECONDARY OUTCOMES:
Change in Mood | 27 weeks
  individual change between initial and final Hamilton Depression Scale (HAMD) score. This will also enable to use the secondary outcome as a covariate of the primary outcome variable
Change in Cognition | 27 weeks
  Alzheimer's Disease Assessment Scale - Cognition (ADAS-Cog)
Deterioration in Cognition | 27 weeks
  Delirium Rating Scale-Revised-98 (DRS-R98)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Sartorius, MD, PhD, Principal Investigator — Department of Psychiatry and Psychotherapy, Central Institute of Mental Health (CIMH), Medical Faculty Mannheim, University of Heidelberg